CLINICAL TRIAL: NCT06409702
Title: A Single-arm Prospective Study of the Treatment in High-risk Newly Diagnosed Multiple Myeloma With Minimal Residual Disease Detection
Brief Title: Treatment of High-risk Newly Diagnosed Multiple Myeloma With Minimal Residual Disease Detection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Fu chengcheng PhD, Deputy Director, Department of Hematology, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKRD-MM11
Record Dates: First submitted 2024-04-16; First posted 2024-05-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Newly Diagnosed; High Risk; MRD; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DKRd (Experimental): All patients will be treated with VRD induction for first-cycle,and then DKRD induction and consolidation therapy for following 5~7 cycles, then maintenance therapy.
  Interventions: Drug: Carfilzomib; Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone; Drug: VRD for first-cycle induction therapy

INTERVENTIONS:
Drug: Carfilzomib — Induction:
  ASCT：20mg/56mg/m2 ,D1,8,15，C2-4; non ASCT: 20mg/36mg/m2 ,D1,8,15，C2-4;
  Consolidation:
  ASCT: 56mg/m2 ,D1,8,15，C5-6; non ASCT: 36mg/m2 ,D1,8,15，C5-8;
  Maintenance:
  ASCT: 70mg/m2 ，D1，15; non-ASCT：56mg/m2 ，D1，15 After consolidation therapy, if MRD negativity is sustained for more than 1 year, carfilzomib will be discontinued
  Other Names: Kyprolis
Drug: Daratumumab — 28d/Cycle
  Induction:
  16mg/kg, D1,8,15,22，C 2-3，16mg/kg, D1,15, C4;
  Consolidation:
  ASCT: 16mg/kg/d, D1,15,C5-6; non ASCT: 16mg/kg/d, D1,15,C5-8;
  Maintenance:
  16mg/kg, D1,monthly After consolidation therapy, if MRD negativity is sustained for more than 1 year, daratumumab will be discontinued
  Other Names: Darzalex
Drug: Lenalidomide — 28d/Cycle
  Induction:
  25mg qd d1-21 C2-C4;
  Consolidation:
  ASCT: 10mg d1-21，C5-6; non ASCT: 25 mg d1-21，C5-8;
  Maintenance: 10mgqd D1-21
  After consolidation therapy, if MRD negativity is sustained for more than 1 year, lenalidomide monotherapy will be maintained until disease progression
Drug: Dexamethasone — 28d/Cycle
  Induction:
  ASCT：40mg qd, po/iv，D1,8,15,22，C2-4; non ASCT:20mg qd, po/iv，D1,8,15,22，C2-4;
  Consolidation:
  ASCT: 40mg qd, po/iv，D1,8,15,22，C5-6; non ASCT:20mg qd, po/iv，D1,8,15,22，C5-8
Drug: VRD for first-cycle induction therapy — Induction:
  C1, 28d/cycle Bortezomib(V）:1.3 mg/m2，H，d1、4、8、11； Lenalidomide(R)：25mg，po. qd d1-14; Dexamethasone(D)：20 mg，po/iv，D1，2, 4，5, 8，9, 11,12。
  Other Names: Bortezomib(V), Lenalidomide(R), Dexamethasone(D)

SUMMARY:
The goal of this study is to evaluate sustained MRD negativity for one year in DKRD induction & consolidation therapy +/- ASCT in newly diagnosed high-risk multiple myeloma patients. It aims to evaluate the efficacy and safety of the combination regimen of Daratumumab in combination with carfilzomib, lenalidomide, and dexamethasone (DKRD) +/- ASCT for the treatment of patients with newly diagnosed high-risk multiple myeloma. Participants will receive bortezomib based induction therapy for one cycle, and then DKRD induction for 3 cycles(+ASCT), DKRD consolidation for 2-4 cycles, and DKR maintenance treatment(adjusted according to MRD negativity after consolidation therapy)

DETAILED DESCRIPTION:
Daratumumab, carfilzomib, lenalidomide and dexamethasone are commonly used drugs for multiple myeloma. The efficacy of their combination has been proven in newly diagnosed multiple myeloma patients, including high-risk patients, while there are no relevant data in the Chinese population. Therefore, the efficacy of DKRd regimen in Chinese HR-NDMM patients needs to be further explored.

It is a prospective, single-arm study. High risk(HR)-NDMM Patients with will be recruited and their baseline data will be collected. Patients will be treated with bortezomib, lenalidomide and dexamethasone for the first cycle in order to urgently relieve bone pain, renal insufficiency, hypercalcemia and other symptoms, during which screening and evaluation is conducted. And then patients will be treated with 3 cycles of daratumumab, carfilzomib (K) lenalidomide (R) combined with dexamethasone (d), after which stem cells were collected from transplant-eligible, followed by autologous hematopoietic stem cell transplantation, two cycles of DKRD consolidation, DKR maintenance treatment for more than one year. If continuous MRD negativity for more than one year, patients will be treated with only lenalidomide maintenance. Transplant-noneligible patients will be treated with DKRD for 4-cycles consolidation therapy without transplantation, and then entered DKR maintenance therapy. If patients with continuous MRD negativity for more than one year will be treated with only lenalidomide maintenance. Follow-up was conducted and outcome indicators were collected to explore the efficacy and safety of DKRd treatment in HR-NDMM patients. The results of this study are expected to provide new treatment options and corresponding dosages for Chinese HR-NDMM patients, thereby improving patient outcomes and reducing the overall disease burden.

ELIGIBILITY:
Inclusion Criteria:

1. patients with newly diagnosed multiple myeloma（may receive up to one course of a bortezomib-containing regimen for the urgent relief of bone pain, renal insufficiency, and hypercalcemia）;
2. age ≥ 18 years;
3. have an evaluable lesion; serum M protein ≥ 10 g/L, or urinary light chain ≥ 200 mg/24h, or involved serum free light chain (FLC) ≥ 100 mg/L, and an extramedullary measurable tumor SPD: The diameter of cutaneous nodules can be measured with a manual tape, and extramedullary tumor SPD of extramedullary tumors is measured on a CT scan as the product of the largest dimension of the largest pendulous diameter of the lesion (minimum diameter of 5mm or more), parosteal lesions need to be in soft tissue outside the bone cavity to meet the above criteria. MRI measures the size of an extramedullary tumor as the product of the maximum pendulous diameter at the level of the largest area of the tumor (minimum diameter of 5mm or more)
4. ECOG physical status score ≤ 2
5. or have a high-risk karyotype abnormality recognized in mSMART or NCCN guidelines: t(4;14), t(14;16), t(14;20), Del(17p) or -17 and/or TP53 mutation, Del(1p32), 1q21 gain(amp), the coexistence of two adverse karyotypes as a double hit,and triple hit similarly defined
6. or R-ISS stage 3
7. or combined plasma cell leukemia (defined as peripheral blood sorted clonal plasma cells ≥ 5%)
8. bone marrow function: neutrophils ≥ 1.0 x 109 /L, platelets ≥ 70 x 109 /L (if bone marrow plasma cells ≥ 50%, platelets ≥ 50 x 109 /L)
9. AST, ALT, ALP ≤ 3 × upper limit of normal value, serum bilirubin ≤ 2 times upper limit of normal value;
10. serum creatinine clearance ≥ 40mL/min
11. negative pregnancy test for women of childbearing age; patients and their spouses must agree to use effective contraception during the treatment period and the following one-year period;
12. Signed informed consent for chemotherapy. A legal representative will sign the informed consent form if the subject is unable to sign it due to impaired consciousness, paralysis of the subject's upper limbs, or inability to write.

Exclusion Criteria:

1. monoclonal gammopathy of undetermined significance (MGUS), smoldering myeloma, primary light chain amyloidosis with organ involvement.
2. diagnosed or treated for another malignancy prior to pre-registration ≤ 1 year or previously diagnosed with another malignancy with evidence of any residual disease being treated.
3. other co-morbidities that would interfere with the subject's ability to participate in the trial, e.g., uncontrolled infections, uncompensated cardiac or pulmonary disease, other synchronized chemotherapy or any adjuvant therapy considered investigational.
4. peripheral neuropathy ≥ grade 1-2 with pain on clinical examination within 30 days prior to pre-registration
5. major surgery within 14 days prior to pre-registration
6. evidence of current uncontrolled cardiovascular disease, including uncontrolled hypertension (hypertension defined as SBP ≥ 140 mmHg and/or DBP ≥ 90 mmHg on 3 non-same day office measurements without antihypertensive medication), arrhythmias (prolonged QT interval, ventricular tachycardia, ventricular flutter, ventricular fibrillation, frequent ventricular premature beats (24 h ventricular premature load ≥ 15% of the total number of heart beats, atrioventricular block, heart rate <30-40 bpm), congestive heart failure, unstable angina or myocardial infarction. New York Heart Association (NYHA) Class III, IV heart failure.
7. Participants with known chronic obstructive pulmonary disease (COPD) (defined as exertional expiratory volume in 1 second [FEV1] <50% of predicted normal volume), persistent asthma, or a history of asthma within the past 2 years (controlled intermittent asthma or mild persistent asthma is permitted). Participants with known or suspected COPD must have FEV1 testing during screening.
8. moderate/severe renal insufficiency: creatinine clearance < 40mL/min.
9. known human immunodeficiency virus (HIV) positivity.
10. Hepatitis B seropositivity (defined as a positive Hepatitis B surface antigen [HBsAg] test). Subjects whose infection has resolved (i.e., subjects who are HBsAg negative but positive for Hepatitis B Core Antigen Antibody [anti-HBc] and/or Hepatitis B Surface Antigen Antibody [anti-HBs]) must be screened for Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) levels using real-time Polymerase Chain Reaction (PCR). PCR-positive subjects will be excluded. Exception:Subjects with serologic results suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) and a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.
11. known or suspected active hepatitis C infection.
12. any medical or psychiatric condition that, in the opinion of the investigator, may interfere with the completion of treatment under this protocol.
13. known allergy or intolerance to the test drug.
14. inability to comply with the protocol/procedure.
15. Subjects will be ineligible to participate in the trial because the genotoxic, mutagenic, and teratogenic effects of the investigational drug(s) involved in this trial on the developing fetus and neonate are unknown if any of the following conditions are present at the time of screening: Pregnant women, lactating mothers, males or females of childbearing potential who refuse adequate contraception (as per protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MRD negative rate | Completion of consolidation therapy
  the rate of minimal residual disease negativity

SECONDARY OUTCOMES:
≥VGPR rate | after completion of induction therapy (about 4 months after enrollment) and consolidation therapy(about 11 months after enrollment) , respectively
  the rate of very good partial response or better
overall response rate | after completion of induction therapy (about 4 months after enrollment) and consolidation therapy(about 11 months after enrollment) , respectively
  the rate pf overall response
adverse events | from enrollment to completion of following up, about 2 years
  the rate of adverse events and grade of adverse events
PFS | from enrollment to completion of one-year maintenance therapy
  Progression-free survival
OS | from enrollment to completion of one-year maintenance therapy
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China